CLINICAL TRIAL: NCT00636389
Title: Urea, Phosphate and b2-Microglobulin Removal and Ease of Use: Comparing the Polyflux HD-C4 With the Polyflux 210H
Brief Title: Molecule Removal and Ease of Use: A Comparison of Two Different Dialyzers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Gambro Renal Products, Inc. (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Gambro 1460
Record Dates: First submitted 2008-02-13; First posted 2008-03-14 (Estimated); Results first posted 2011-08-11 (Estimated); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Disease
Keywords: Hemodialysis; Dialysis, Renal; Dialysis, Extracorporeal; Extracorporeal Dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HD-C4 First, then 210H (Other): Subjects will be randomly assigned to begin the first week of three consecutive treatments with the Polyflux HD-C4 dialyzer. Following the third treatment, the subjects will be switched to the Polyflux 210H dialyzer for a second week of three consecutive treatments. Therefore each subject will have a total of six consecutive dialysis treatments.
  Interventions: Device: Polyflux 210H dialyzer; Device: Polyflux HD-C4
- 210H First, then HD-C4 (Other): Subjects will be randomly assigned to begin the first week of three consecutive treatments with the Polyflux 210H dialyzer. Following the third treatment, the subjects will be switched to the Polyflux HD-C4 dialyzer for a second week of three consecutive treatments. Therefore each subject will have a total of six consecutive dialysis treatments.
  Interventions: Device: Polyflux 210H dialyzer; Device: Polyflux HD-C4

INTERVENTIONS:
Device: Polyflux 210H dialyzer — Three consecutive treatments with the Polyflux 210H dialyzer. All study treatments will be performed in the standard hemodialysis mode.
  Other Names: Gambro Polyflux 210H dialyzer
Device: Polyflux HD-C4 — Three consecutive treatments with the Polyflux HD-C4 dialyzer. All study treatments will be performed in the standard hemodialysis mode.
  Other Names: Gambro Revaclear

SUMMARY:
The Polyflux HD-C4 (Gambro Renal Products) is a new dialyzer based on the existing Polyflux H membrane and dialyzer technology, but which achieves a performance comparable to Polyflux 210H in a significantly smaller device.

The objectives of this study are:

1. To compare and contrast small and large molecule removal by the Polyflux HD-C4 and Polyflux 210H dialyzers under conditions of routine hemodialysis; and,
2. To compare and contrast the ease of use of the Polyflux HD-C4 dialyzer with that of the Polyflux 210H under conditions of routine clinical use for hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* Stable hemodialysis prescription using Polyflux 210H or Polyflux 21R for at least 2 months prior to study enrollment
* Dialyzing through a native fistula or Gore-Tex graft.
* Blood access must be able to provide a blood flow rate of 400 ml/min.

Exclusion Criteria:

* Non-compliance with dialysis
* Hematocrit less than 28%
* Active Infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry Alcorn Jr., PharmD, Principal Investigator — Davita Clinical Research Facility
Locations (1):
- DaVita Clinical Research Facility, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Daugirdas JT. Second generation logarithmic estimates of single-pool variable volume Kt/V: an analysis of error. J Am Soc Nephrol. 1993 Nov;4(5):1205-13. doi: 10.1681/ASN.V451205. PMID 8305648
- [Background] Daugirdas JT, Schneditz D. Overestimation of hemodialysis dose depends on dialysis efficiency by regional blood flow but not by conventional two pool urea kinetic analysis. ASAIO J. 1995 Jul-Sep;41(3):M719-24. doi: 10.1097/00002480-199507000-00107. PMID 8573901

RESULTS

PARTICIPANT FLOW:
Groups:
- HD-C4 First (Period 1), Then 210H (Period 2): Subjects were randomly assigned to begin the first week (Period 1) of three consecutive treatments with the Polyflux HD-C4 dialyzer. Following the third treatment, the subjects were switched to the Polyflux 210H dialyzer for a second week (Period 2) of three consecutive treatments. Therefore each subject had a total of six consecutive dialysis treatments.
- 210H First (Period 1), Then HD-C4 (Period 2): Subjects were randomly assigned to begin the first week (Period 1)of three consecutive treatments with the Polyflux 210H dialyzer. Following the third treatment, the subjects were switched to the Polyflux HD-C4 dialyzer for a second week (Period 2) of three consecutive treatments. Therefore each subject had a total of six consecutive dialysis treatments.
Period: Period 1 - 1 Week
Arm/Group | HD-C4 First (Period 1), Then 210H (Period 2) | 210H First (Period 1), Then HD-C4 (Period 2)
Started | 7 | 5
Completed | 7 | 5
Not Completed | 0 | 0
Period: Period 2 - 1 Week
Arm/Group | HD-C4 First (Period 1), Then 210H (Period 2) | 210H First (Period 1), Then HD-C4 (Period 2)
Started | 7 | 5
Completed | 7 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Urea Removal Under Conditions of Routine Hemodialysis.
Description: Urea removal is correlated with successful clinical outcomes. Kt/V is a way of measuring the delivered dose of dialysis where K=clearance of urea, t=treatment time and V=volume of body water. Single-pool (sp) Kt/V assumes that urea is removed from a single compartment in the human body during dialysis. However, because there are multiple compartments in the human body, rebound occurs following hemodialysis which lowers the Kt/V. Equilibrated (e) Kt/V is an equation that has been devised to predict the amount of rebound based on the ratio of K/V. Outcomes are posted for both spKt/V and eKt/V.
Time Frame: 2 weeks = duration required for each subject to complete 6 consecutive dialysis treatments
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | HD-C4 | 210H
Number analyzed (Participants) | 12 | 12
ratio
  Single-pool Kt/V Urea | 1.64 (0.26) | 1.61 (0.24)
  Equilibrated Kt/V | 1.42 (0.22) | 1.40 (0.22)

2. Secondary Outcome: Comparison of Dialyzer Ease of Use Between the Polyflux HD-C4 Dialyzer and the Polyflux 210H
Description: Assessment of blood side priming: 1=Very Easy 2=Acceptable 3=Difficult 4=Very Difficult / Assessment of dialysate side priming: 1=Perfect 2=Acceptable 3= Not Acceptable / Appearance of dialyzer fibers: 1=Very Good 2=Good 3=Poor 4=Very Poor / Appearance of dialyzer arterial header: 1=Very Good 2=Good 3=Poor 4=Very Poor / Appearance of venous header: 1=Very Good 2=Good 3=Poor 4=Very Poor /
Time Frame: 2 weeks = duration required for each subject to complete 6 consecutive dialysis treatments
Population: Each of the 12 subjects underwent three consecutive treatments with the HD-C4 and three consecutive treatments with the Polyflux 210H.
Measure: Mean (Standard Deviation); unit: Units on a Scale 1 = Best
Units Other Than Participants: dialyzers
Arm/Group | HD-C4 | 210H
Number analyzed (Participants) | 12 | 12
Number analyzed (dialyzers) | 36 | 36
Units on a Scale 1 = Best
  Priming of blood compartment | 1.19 (0.40) | 1.47 (0.51)
  Priming of dialysate compartment | 1.36 (0.49) | 1.51 (0.51)
  Appearance of fibers | 1.42 (0.55) | 1.78 (0.64)
  Appearance of arterial header | 1.61 (0.55) | 1.72 (0.51)
  Appearance of venous header | 1.57 (0.74) | 1.77 (0.55)

3. Primary Outcome: A Comparison of Pre- to Post-dialysis Reduction of Small and Large Molecules Under Conditions of Routine Hemodialysis.
Description: Overall removal of urea, phosphorus and β2-microglobulin was determined from the pre- to post-dialysis change in plasma concentration and from the amount of solute recovered in the dialysate. This outcome measure is reported as the percentage of pre- to post-dialysis reduction of urea, phosphorus and β2-microglobulin.
Time Frame: 2 weeks = duration required for each subject to complete 6 consecutive dialysis treatments
Measure: Mean (Standard Deviation); unit: Percentage of reduction
Arm/Group | HD-C4 | 210H
Number analyzed (Participants) | 12 | 12
Percentage of reduction
  Urea Pre- to post-dialysis reduction (%) | 74 (6) | 74 (5)
  Phosphorus Pre- to post-dialysis reduction (%) | 61 (9) | 60 (17)
  b2-microglobulin Pre- to post-dialysis reduct (%) | 52 (12) | 58 (8)

ADVERSE EVENTS:
Time Frame: 1 year, 1 month
Arm/Group | HD-C4 First (Period 1), Then 210H (Period 2) | 210H First (Period 1), Then HD-C4 (Period 2)
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 0/7 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days